CLINICAL TRIAL: NCT03410355
Title: The Use of Bone Marrow Aspirate Concentrate in the Context of Hip Osteoarthritis: A Randomized Controlled Trial
Brief Title: Bone Marrow Aspirate Concentrate Use in Hip Osteoarthritis
Acronym: BMAC
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Health Canada no longer allowed use of BMAC
Sponsor: Nova Scotia Health Authority (Other)
Responsible Party: Principal Investigator, Ivan Wong, Orthopaedic Surgeon MD FRCS(C), Dip. Sports Medicine, Nova Scotia Health Authority
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IW-001
Record Dates: First submitted 2017-12-22; First posted 2018-01-25 (Actual); Last update posted 2022-03-08 (Actual); Status verified 2022-03

CONDITIONS: Osteoarthritis, Hip
MeSH Terms: conditions — Osteoarthritis, Hip | interventions — Cortisone

STUDY DESIGN:
Intervention Model Description: randomized control trial
Who Masked: Outcomes Assessor
Masking Description: The outcomes assessor will be blinded to the intervention
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- BMAC/PRP Injection Group (Experimental): This group will receive an injection of BMAC/PRP for treatment of OA
  Interventions: Procedure: BMAC/PRP Injection
- Cortisone Injection Group (Active Comparator): This group will receive an injection of cortisone for treatment of OA
  Interventions: Procedure: Cortisone Injection

INTERVENTIONS:
Procedure: BMAC/PRP Injection — Patients will be placed on an office procedure under local anesthesia. The investigators will harvest 60 cm3 of bone marrow from posterior iliac crest and centrifuged obtaining approximately 3 cm3 of autologous bone marrow-mesenchymal stem cells concentrate. At the same time, 60cm3 of peripheral blood will be taken and centrifugated once, to obtain approximately 3 cm3 of PRP. After activation of platelet rich plasma cells they will be mixed in one syringe with the concentrated BMaC and both will be injected in the hip joint under ultrasound.
  Arms: BMAC/PRP Injection Group
Procedure: Cortisone Injection — An intraarticular injection of 1cm3 with 80mg of methylprednisolone combined with 3cm3 of 0.25% bupivacaine will be injected in the hip joint under ultrasound.
  Arms: Cortisone Injection Group

SUMMARY:
The purpose of this study is to evaluate the effect of combined Bone marrow aspirate concentrate (BMAC) and Platelet Rich Plasma (PRP) action after a single hip intraarticular injection to young symptomatic patients with primary radiologic stage of hip OA (Kellgren-Lawrence grade I or II) compared to a control local anesthetic with cortisone injection group of patients. The hypothesis is that the patients with hip OA will benefit more and for longer from OA symptoms in the BMAC and PRP group rather than in the group of local anaesthetic and cortisone. Furthermore, this study could be valuable in determining the safety and effectiveness of the BMAC and PRP combined injection for early low grade hip OA in young active patients who are neither good candidates for total hip replacement nor preservative hip surgery.

DETAILED DESCRIPTION:
The protocol will be applied to a blinded randomized controlled study. Patients who fit the inclusion criteria and have consented to the trial, will be randomized to receive a single injection of BMAC with PRP or local anesthetic with cortisone.

Pre-Injection Procedures:

Patients will receive a clinical evaluation where they will complete the HHS, the WOMAC score, the VR-12 form, VAS score, and the two functional assessment tests to assess pain and function prior to the injection. The two functional assessments will be performed by the blinded researcher. Following the evaluation, the patients will receive an intra-articular hip injection.

Injection Procedures:

Control group: In the second group of patients, an intraarticular injection of 1cm3 with 80mg of methylprednisolone combined with 3cm3 of 0.25% bupivacaine will be performed in the same manner with the first group.

Experimental group: In the first group, patients will be placed on an office procedure under local anesthesia. The investigators will harvest 60 cm3 of bone marrow from posterior iliac crest and centrifuged obtaining approximately 3 cm3 of autologous bone marrow-mesenchymal stem cells concentrate. At the same time, 60cm3 of peripheral blood will be taken and centrifugated once, to obtain approximately 3 cm3 of PRP. After activation of platelet rich plasma cells they will be mixed in one syringe with the concentrated BMaC and both will be injected in the hip joint under ultrasound. In all cases four samples of 0.2cm3 will be collected, one with patient's whole blood, one with the PRPs final mixture, one with whole bone marrow aspirate, and one with the BMaCs final mixture, and will be sent to the NSHA Hematology Laboratory for cell quantification. The leukocyte counts and differential (neutrophils, monocytes, lymphocytes, eosinophils and basophils) as well as thrombocyte counts in all samples will be determined using Automated Hematology Analyzer (Sysmex). Percentages of mature and immature leukocytes in the bone marrow aspirate and BMaC samples will be determined by standard morphologic examination using slides prepared with the Wright's stain. CD34+ stem cell enumeration in the bone marrow aspirate sample and BMaC will be performed by flow cytometry (Canto II Analyser).The concentration factor of PRP will be calculated from the quotient of the thrombocyte count in whole blood and in PRP. Additionally, IGF-I, VEGF, TGF-b, bFGF, HGF and PDGF will be quantified in serum or plasma and in PRP using commercially available ELISA kits (QuantikineH, ELISA KITS, R&D Systems, USA).

Post-Injection Procedures:

Clinic visits will occur at 6, 12, 24, and 48 weeks post-injection to perform clinical evaluations with outcome measures of the patients. All collected data will be statistically analyzed to check the effect of BMAC and PRP intraarticular hip injections in young patients with early OA. The investigators will also document the activity level of all participants (type of sport or activity participated in and the intensity and volume of participation) and correlate it with the outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Age <60 years old
* BMI of <40 kg/m2
* Able to walk 50m unaided and not confined to a wheel chair
* Unilateral hip pain and radiographically and arthroscopically verified OA of the hip within the last 6 months (Kellgren-Lawrence grade I or II)
* HHS of less than 80
* Ability to understand the informed consent and participation instructions Attempted to use over the counter therapy without relief
* Able to participate for the entire protocol study period
* Able to follow physicians directions

Exclusion Criteria:

* Clinically significant OA in the contralateral hip
* Clinically significant pain in any other joint
* Have had intra-articular BMAC and or PRP injection within the preceding six months in the study hip
* Have had intra-articular steroid injection within the preceding three months in the study hip
* Have had previous surgical procedures on the affected hip within the preceding 6 months
* Have had a serious injury to the study hip within the previous 3 months
* Have had a serious psychological or medical condition that would interfere with their involvement
* Have had treatment with pain medications other than Tylenol and the drug remains in their system at the baseline or first study visit
* Have used of opioids other than weak opioids for OA pain more than 3 days/week within the last month
* Have used of systemic glucocorticoids (excluding inhaled steroids) within the preceding 3 months
* Treatment started with glucosamine/chondroitin sulfate or if the dosing has not been stable in the previous three months
* Has had a history of septic arthritis, skin infection or disease in the region of the injection site
* Currently using an anticoagulant excluding Aspirin 325 mg/day
* Uncontrolled diabetes
* Has any medical condition the principal investigator believes deems the patient unsuitable for the study
* Has any pathology of lumbar spine, sacroiliac (SI) joints, neuropathic or extra-articular hip pain
* Has a history of alcohol or drug abuse within the six months prior to enrolment in the study
* Has had a diagnosis of rheumatoid arthritis
* Has had a diagnosis of ankylosing spondylitis
* Has had a diagnosis of psoriatic arthritis
* Has had a diagnosis of reactive arthritis
* Has had a diagnosis of gout
* Has had a diagnosis of any connective tissue disease.

Ages: 16 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 6 (Actual)
Dates: Start 2018-02-01 (Actual); Primary Completion 2019-05-17 (Actual); Study Completion 2019-05-17 (Actual)

PRIMARY OUTCOMES:
Functional Benefit and Pain Level Changes using iHOT33 Questionnaire | 6 months
  Assessment of functional benefit and pain level changes, using the International Hip Outcome Tool (iHot33) score at the 6-month time point post-injection, as well as, the pre-injection iHot33 score. The iHOT33 is a 33 question tool used to assess a patients ability to return to an active lifestyle through a subjective measurement of symptoms as well as emotional and social health status. Patients use a visual analog type scale (VAS) for each of the 33 questions to determine if activities are extremely difficult (to the left) to not difficult at all (to the right). Score is calculated as a mean on all VAS scores measured in millimeters, with 100 being the best score and 0 being the worst.

SECONDARY OUTCOMES:
Functional Benefit and Pain level Changes using the modified Harris Hip Score (HHS) | 6 months
  The HHS is a widely used 10 item evaluation used to assess hip pain, function, hip deformity, and range of motion in patients who have total hip replacements, femoral neck fractures, and osteoarthritis. Each question is assigned a different numerical value. A score of 90-100 is excellent indicating minimal pain and excellent function, 80-89 is good, 70-79 fair, 60-69 poor, and below 60 a failed result.
Functional Benefit and Pain level Changes using the The Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) | 6 months
  The WOMAC is a 24 item evaluation used in hip or knee OA to assess pain, stiffness, and physical function. This questionnaire measures five items for pain (score range 0-20), two for stiffness (score range 0-8), and 17 for functional limitation (score range 0-68). All questions ask participants to report their level of difficulty performing different tasks, 0 = None, 1 = Slight, 2 = Moderate, 3 = Very, 4 = Extremely. The score is calculated as a percentage of 96. With 100% being the worst and 0% being the best.
Burden of Disease and Quality of Life Changes using the Veterans RAND 12 Item Health Survey (VR-12) | 6 months
  This instrument is primarily used to measure health related quality of life, to estimate disease burden and to evaluate disease-specific impact on general and selected populations. The items on the questionnaire correspond to eight principal health domains including general health perceptions, physical functioning, role limitations due to physical and emotional problems, bodily pain, energy-fatigue, social functioning, and mental health.
Pain Changes using the Visual Analogue Scale (VAS) | 6 months
  The VAS is the most common pain scale for quantification of disease related pain.This consists of a horizontal line, 100 mm in length, anchored by word descriptors at each end, "no pain" and "very severe pain" respectively. The patient marks on the line the point that they feel represents their perception of their current state. The VAS score is determined by measuring in millimeters from the left-hand end of the line to the point that the patient marks. 100 mm=very severe pain, 0mm=no pain.

CONTACTS AND LOCATIONS:
Overall Officials: Ivan Wong, MD, Principal Investigator — Nova Scotia Health Authority
Locations (1):
- Nova Scotia Health Authority, Halifax, Nova Scotia, Canada

IPD SHARING:
Plan to Share IPD: Undecided